CLINICAL TRIAL: NCT04652778
Title: Safety & Performance of Ablation With the Centauri System for the Elimination of Atrial Fibrillation (SPACE AF)
Brief Title: Safety & Performance of the Centauri System for Patients With Atrial Fibrillation
Acronym: SPACE AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Galaxy Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-00008
Record Dates: First submitted 2020-11-20; First posted 2020-12-03 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Pulsed Field Ablation (PFA) using the Centauri System

INTERVENTIONS:
Device: Pulsed Field Ablation (PFA) using the Centauri System — cardiac ablation using pulsed electric field energy to cause pulmonary vein isolation; cavo-tricuspid isthmus (CTI) line ablation may be performed as needed

SUMMARY:
This is a prospective, single-arm, open-label clinical study following patients to 1 year, to evaluate the safety and performance of the Centauri system for catheter ablation of atrial fibrillation (AF). The study will include adult patients (age 18-75 years) who are indicated for a first-time catheter ablation of AF where the pre-procedure treatment plan contemplates pulmonary vein isolation (PVI) in patients with paroxysmal AF (PAF), and PVI - with or without additional left atrial ablations - in patients with Persistent AF (PeAF) of short duration (< 1 year).

ELIGIBILITY:
Inclusion Criteria:

1. Failure of at least one antiarrhythmic drug (AAD) (Class I - IV) for AF, as evidenced by recurrent symptomatic AF or intolerable side effects due to AAD
2. Diagnosis of recurrent symptomatic paroxysmal AF (PAF) or short duration (< 1 year) Persistent AF (PeAF) with the following documentation:

   a. PAF i. Physician's note indicating symptoms consistent with recurrent symptomatic PAF AND ii. ≥ 2 episodes of PAF within 12 months prior to enrollment. At least one episode should be documented by ECG, transtelephonic monitor (TTM), Holter monitor, telemetry strip or similar, showing at least 30 seconds of AF b. PeAF i. Physician's note indicating symptoms consistent with continuous AF episode lasting longer than 7 days but less than 1 year AND ii. Any 24-hour continuous ECG recording documenting persistent AF within 6 months prior to enrollment OR iii. Two ECGs from any form of rhythm monitoring showing continuous AF taken at least 7 days apart within 12 months prior to enrollment OR iv. History of direct current cardioversion (DCCV) performed within 12 months prior to enrollment
3. Age 18 through 75 years-old on the day of enrollment
4. Patient is indicated for an ablation procedure according to society guidelines or investigational site practice
5. Patient is willing and able to give informed consent.
6. Patient is willing, able, and committed to participate in baseline and follow-up evaluations for the full duration of the study.

Exclusion Criteria:

1. Long-standing persistent AF (continuous AF sustained > 1 year)
2. AF secondary to electrolyte imbalance, thyroid disease, alcohol abuse, or other reversible/non-cardiac causes
3. Left atrial anteroposterior diameter > 5.0 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT) within 6 months prior to enrollment
4. Patient who is not on oral anticoagulation therapy for at least 3 weeks prior to the index ablation procedure
5. Use of amiodarone within 6 weeks prior to enrollment
6. Prior left atrial ablation or surgical procedure (including left atrial appendage (LAA) device or occlusion)
7. Planned LAA closure procedure or implant of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function) for any time during the follow-up period
8. Presence of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
9. Presence of any pulmonary vein stents
10. Presence of any pre-existing pulmonary vein stenosis
11. Pre-existing hemidiaphragmatic paralysis
12. Atrial or ventricular septal defect closure
13. Atrial myxoma
14. Presence of any prosthetic heart valve
15. Hemodynamically significant valvular disease
16. History of pericarditis
17. History of Rheumatic heart disease
18. History of thromboembolic event within 6 months of time of enrollment or evidence of intracardiac thrombus at time of procedure
19. Any of the following events within 3 months of enrollment

    * Myocardial infarction (MI)
    * Unstable angina
    * Percutaneous coronary intervention
    * Heart surgery including coronary artery bypass grafting
    * Heart failure hospitalization
    * Cerebral ischemic event (stroke or transient ischemic attack (TIA))

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Device and Procedure related serious adverse event rate | 30 days
  The rate of system-related and procedure-related serious adverse events of interest
Acute Procedural Success | During treatment procedure
  Proportion of patients with confirmed pulmonary vein isolation (PVI) during the index procedure
Chronic Success | 12 months
  Proportion of patients with freedom from AF recurrence after a single procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada